CLINICAL TRIAL: NCT05934435
Title: Addressing Pain Care Inequities With Empowered Relief Delivered by ASPMN Nurses: A Randomized Controlled Trial
Brief Title: Empowered Relief Delivered by Nurses
Acronym: ERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: American Society for Pain Management Nursing (Unknown)
Responsible Party: Principal Investigator, Marian Wilson, Associate Professor, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20013-001
Record Dates: First submitted 2023-06-17; First posted 2023-07-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Pain, Chronic
Keywords: Pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: After randomized 1:1 to one of two unblinded study groups: ER and Wait-List Control, participants randomized to the ER group will complete the ER class. A crossover intervention class will be offered to those patient participants randomized to WLC once the ER group has completed their class and follow up assessments, estimated at 2 months post intervention.
Who Masked: Outcomes Assessor
Masking Description: Biostatistician will be blinded to ER treatment group or Wait-list Control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empowered Relief treatment (Experimental): Participants randomized to the ER group will complete a HIPAA compliant, password protected 2-hour Zoom ER class delivered by an ER-trained ASPMN nurse.
  Interventions: Other: Empowered Relief
- Wait-list Control (Other): Participants randomized to the Wait-list Control group will continue their usual pain care for 2 months and complete surveys to compare with the experimental treatment group. After serving as controls, they will be invited to attend the 2-hour Zoom ER class delivered by an ER-trained ASPMN nurse.
  Interventions: Other: Empowered Relief

INTERVENTIONS:
Other: Empowered Relief — psycho-educational pain skills training
  Other Names: ER

SUMMARY:
This study will investigate effects of a psychoeducation pain management skills intervention on adults with persistent pain by training a cohort of American Society for Pain Management Nursing (ASPMN) nurses to deliver and it [Empowered Relief (ER)], as a single-session video-conferenced program. The primary objective is to evaluate the effects of ASPMN nurse-provided ER versus waitlist control (WLC) on pain catastrophizing, pain bothersomeness, pain intensity, pain interference, sleep disturbance, physical function, depression, anxiety, and social isolation for patients with persistent pain. Secondarily, feasibility and acceptability of the ER program will be assessed through recruitment and retention data and qualitative satisfaction data.

DETAILED DESCRIPTION:
Design: This study will be conducted as a randomized controlled trial comparing effects of ER to a WLC of participants with persistent pain when ER is provided by ER-trained ASPMN nurses. The secondary aims of feasibility and acceptability will use qualitative descriptive methods.

Participants: Participants (N=170) will be adults aged 18 and above years with self- reported or clinically diagnosed persistent pain. Participants will be recruited at clinical sites identified by ER-trained nurses and can be self or clinician referred. Participants will complete an online eligibility form to screen for inclusion and exclusion criteria. Inclusion criteria: pain >3 months more than half the time, English fluency, ability to attend a one-time web-based class and complete web-based surveys, age > 18 years. Exclusion criteria: Previous participation in ER class, cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material or full participation in the study as determined by the investigators.

Procedures: Twenty ASPMN nurses will receive ER training facilitated by Stanford Pain Relief Innovations Lab. ER- trained nurse providers will be ASPMN-member nurses of any clinical background. ASPMN nurses will be invited to apply to become a trainer with the following expectations: ability to fully participate in a live, online, 2-day ER instructor training, able to fluently complete instructor training and deliver the ER program in English, commitment to deliver 1-3 live, online, 2-hour ER programs for patient participants, and willingness to complete post-program surveys after each session they deliver reporting on number of participants and any barriers encountered. Recruitment will occur through ASPMN-related mechanisms of communication, including its website, national officers and directors, newsletter, research group, national committees, chapter leadership and listserv.

After meeting eligibility criteria and completing informed consent, study participants will be asked to complete a baseline survey of demographics and health variables (as outlined in Table 1) and then randomized 1:1 to one of two unblinded study groups: ER and WLC. Participants randomized to the ER group will complete a HIPAA compliant, password protected Zoom ER class delivered by an ER-trained ASPMN nurse. A crossover intervention class will be offered to those patient participants randomized to WLC once the ER group has completed their class and follow up assessments, estimated at 2 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* pain >3 months more than half the time
* English fluency
* ability to attend a one-time web-based class and complete web-based surveys.

Exclusion criteria:

* Previous participation in ER class
* cognitive impairment
* non-English speaking
* psychological factors that would preclude comprehension of material or full participation in the study as determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Change in Pain Catastrophizing | Participants will be assessed at baseline, and then at 2, 4, and 8 week timepoints for change over time.
  Measured by self-report

SECONDARY OUTCOMES:
Change in Pain Intensity | Participants will be assessed at baseline, and then at 2, 4, and 8 week timepoints for change over time.
  0-10 Pain severity scale

CONTACTS AND LOCATIONS:
Overall Officials: Marian Wilson, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Can be requested from principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: Use for secondary analysis